CLINICAL TRIAL: NCT01528462
Title: Does Acute Management of Sleep Disorders Improve Outcomes After Non-disabling Cerebrovascular Events?
Brief Title: Sleep Disorders Managed and Assessed Rapidly in Transient Ischemic Attack (TIA) and In Early Stroke
Acronym: SMARTIES
Status: Completed | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Heart and Stroke Foundation of Canada (Other); Canadian Stroke Network (Other); Sunnybrook Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 277-2011
Record Dates: First submitted 2012-01-03; First posted 2012-02-08 (Estimated); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Stroke; Ischemic Attack, Transient; Sleep Disorders; Sleep Apnea Syndromes; Restless Legs Syndrome
Keywords: Stroke; Ischemic Attack, Transient; Sleep Disorders; Sleep Apnea Syndromes; Restless Legs Syndrome; Chronobiology Disorders
MeSH Terms: conditions — Stroke; Ischemic Attack, Transient; Sleep Wake Disorders; Sleep Apnea Syndromes; Restless Legs Syndrome; Chronobiology Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Expedited Treatment of Sleep Disorders: Please see below.
  Interventions: Other: Expedited Treatment of Sleep Disorders

INTERVENTIONS:
Other: Expedited Treatment of Sleep Disorders — Patients in this arm will undergo an expedited polysomnogram (if clinically necessary) and early treatment of any sleep disorders. Sleep-related disorders will be managed with the currently recommended therapies; patients with obstructive sleep apnea will be treated with positional therapy, continuous positive airway pressure (CPAP), etc., and those with restless legs syndrome will be treated with standard treatments such as iron, or dopaminergic agonists. Patients will also be counselled on improving their sleep hygiene and adjusting the timing of their medication administration to optimize efficacy. Furthermore, patients will receive information handouts.

SUMMARY:
The aim of the investigators was to determine whether the immediate management of any detected sleep disorders can improve outcomes in patients who have had a transient ischemic attack (TIA) or minor stroke. This group of patients is at high risk for having a recurrent stroke or TIA, and the investigators would like to investigate new ways of preventing potentially avoidable events. The treatment of sleep disorders immediately after a stroke or TIA may prove to be a novel method of avoiding future strokes and improving outcomes.

DETAILED DESCRIPTION:
Every year, thousands of people in Canada either die or are permanently disabled after suffering a stroke. This costs our society billions of dollars in physician services, hospital expenses, and decreased productivity. Some individuals are slightly more lucky; instead of having a severe stroke, they have either a very mild stroke or temporary stroke symptoms, also known as a transient ischemic attack (TIA), and do not experience any loss of abilities. However, mild strokes and TIA's can precede the onset of a more serious, disabling stroke. Most of the significant strokes that happen after a mild stroke or TIA occur within days of the original event; there is a need for early interventions that could prevent such occurrences.

One of the goals of recent research has been to find ways to prevent major strokes after individuals have sustained a minor stroke or TIA. Up until now, stroke doctors have focused on treating elevated blood pressures and cholesterol levels, scanning the blood vessels in the neck for significant narrowings, and searching for irregular heart rhythms, all of which are treatable conditions that put patients at risk for having a stroke. Despite research which shows that sleep disorders such as sleep apnea (abnormal pauses in breathing during sleep) or restless legs syndrome (which can cause involuntary leg movements in sleep) are possible risk factors for stroke, these conditions are not routinely investigated by stroke doctors after a TIA or stroke.

The investigators hypothesize that the study patients, who will all receive an expedited sleep assessment and expedited treatment of their sleep disorders, will have at the 3-month follow-up assessment: (i) Significantly improved quality of life at 3 months compared to baseline measurements (primary outcome); (ii) Improved outcomes on measures of sleepiness, psychomotor vigilance, daily function, depressive symptoms, cognition, and blood pressure at 3 months (secondary outcomes).

ELIGIBILITY:
1. Inclusion Criteria:

   * Patients presenting within 14 days of symptoms with either

     * High risk TIA
     * Minor stroke.
   * High risk TIA will be defined as:

     * Transient, acute motor or speech disturbance lasting at least 5 minutes, or
     * Any TIA associated with >50% ipsilateral carotid stenosis (presumed to be symptomatic) or atrial fibrillation not currently anticoagulated
   * Mild stroke will be defined as focal neurological deficits with MRI changes and a National Institutes of Health Stroke Scale score ≤ 5
2. Exclusion Criteria:

   * Past history of impulse control disorder, gambling, or active psychiatric disease
   * Patients with cognitive impairment restricting ability to perform activities of daily function and ability to comply with medical therapy (e.g. CPAP or medication use)
   * Patients with limb weakness not allowing them to utilize a CPAP device
   * Life expectancy less than 6 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Please see eligibility criteria below.
Sampling Method: Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2011-10; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Change in quality of life | Baseline, 3 months
  Quality of life will be measured by the Stroke Specific Quality of Life Scale (Williams LS, Weinberger M, Harris LE, Clark DO, Biller J. Development of a stroke-specific quality of life scale. Stroke 1999;30(7):1362-9).

SECONDARY OUTCOMES:
Change in Epworth Sleepiness Scale | Baseline, 3 months
  The reference for this scale is:
  Johns MW. A new method for measuring daytime sleepiness: the Epworth sleepiness scale. Sleep. 1991 Dec;14(6):540-5.
Change in performance on Psychomotor vigilance task | Baseline, 3 months
  The reference for this measure is:
  Lim J, Dinges DF. Sleep deprivation and vigilant attention. Ann N Y Acad Sci. 2008;1129:305-22.
Change in National Institutes of Health (NIH) Stroke Scale score | Baseline, 3 months
  This is a measure of stroke severity. The reference for this measure is:
  Brott T, Adams HP, Olinger CP, et al. Measurements of acute cerebral infarction: a clinical examination scale. Stroke 1989;July 20(7):864-70.
Change in Barthel Index | Baseline, 3 months
  This scale is used to measure performance in basic activities of daily living. The reference for this measure is:
  Mahoney FI, Barthel D. Functional evaluation: the Barthel Index. Maryland State Medical Journal 1965;14:56-61.
Change in Modified Rankin Scale | Baseline, 3 months
  This scale is used for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke. The reference for this measure is:
  Bonita R, Beaglehole R. Modification of Rankin Scale: Recovery of motor function after stroke. Stroke 1988;19(12):1497-1500.
Change in Montreal Cognitive Assessment (MoCA) score | Baseline, 3 months
  The reference for this measure is: http://www.mocatest.org/
Change in Centre for Epidemiological Studies Depression Scale | Baseline, 3 months
  The reference for this measure is:
  Parikh RM, Eden DT, Price TR, Robinson RG. The sensitivity and specificity of the center for epidemiologic studies depression scale in screening for post-stroke depression. Int J Psychiatry Med. 1988;18:169-181.
Change in serum HgbA1c and fasting lipid profile | Baseline, 3 months
Change in blood pressure | Baseline, 3 months
  Blood pressure will be measured via BpTru Device (www.bptru.com). This device measures the blood pressure 6 times during a single reading; its purpose is to eliminate or reduce the "white coat effect" by discarding the first measurement and averaging the remaining five.

CONTACTS AND LOCATIONS:
Overall Officials: Mark I Boulos, MD MSc, Study Director — Sunybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

REFERENCES:
- [Result] Boulos MI, Murray BJ, Muir RT, Gao F, Szilagyi GM, Huroy M, Kiss A, Walters AS, Black SE, Lim AS, Swartz RH. Periodic Limb Movements and White Matter Hyperintensities in First-Ever Minor Stroke or High-Risk Transient Ischemic Attack. Sleep. 2017 Mar 1;40(3):zsw080. doi: 10.1093/sleep/zsw080. PMID 28329254
- [Result] Dey AK, Alyass A, Muir RT, Black SE, Swartz RH, Murray BJ, Boulos MI. Validity of Self-Report of Cardiovascular Risk Factors in a Population at High Risk for Stroke. J Stroke Cerebrovasc Dis. 2015 Dec;24(12):2860-5. doi: 10.1016/j.jstrokecerebrovasdis.2015.08.022. Epub 2015 Sep 26. PMID 26411693
- [Result] Boulos MI, Wan A, Black SE, Lim AS, Swartz RH, Murray BJ. Restless legs syndrome after high-risk TIA and minor stroke: association with reduced quality of life. Sleep Med. 2017 Sep;37:135-140. doi: 10.1016/j.sleep.2017.05.020. Epub 2017 Jun 30. PMID 28899525
- [Result] Malik PRA, Muir RT, Black SE, Gao F, Swartz RH, Murray BJ, Boulos MI. Subcortical Brain Involvement Is Associated With Impaired Performance on the Psychomotor Vigilance Task After Minor Stroke. Neurorehabil Neural Repair. 2018 Nov;32(11):999-1007. doi: 10.1177/1545968318804415. Epub 2018 Oct 24. PMID 30352529
- [Derived] Veitch MR, AlHamid MA, Muir RT, Dharmakulaseelan L, Ramirez JR, Gao F, Swartz RH, Murray BJ, Black SE, Boulos MI. Association between cerebral small vessel disease and periodic limb movements of sleep in patients with stroke/TIA. Sleep. 2025 Apr 11;48(4):zsaf027. doi: 10.1093/sleep/zsaf027. PMID 39901803